CLINICAL TRIAL: NCT03570073
Title: Prospective Comparative Study of Two Manual and Automated Oocyte Vitrification Systems: Randomization of Mature Oocytes in Vitro of In Vitro Fertilization Attempts With Micro-injection at the "Centre d'Assistance Médicale à la Procréation" of the Dijon University Hospital
Brief Title: Interest of Automated Oocyte Freezing
Acronym: Instruvit
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Centre Hospitalier Universitaire Dijon (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: Barberet AOI 2017
Record Dates: First submitted 2018-06-05; First posted 2018-06-26 (Actual); Last update posted 2018-06-26 (Actual); Status verified 2018-04

CONDITIONS: Automatic Vitrification; Manual Vitrification
MeSH Terms: interventions — Vitrification

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Manual vitrification (Active Comparator)
  Interventions: Other: Manual vitrification
- Automatic vitrification (Experimental)
  Interventions: Other: Vitrification with GaviTM system

INTERVENTIONS:
Other: Manual vitrification — Two oocytes will be frozen by vitrification. At thawing, the degree of rehydration objectified by the measurement of oocyte surfaces and the appearance of potential lysis will be studied thanks to culture in the embryoscope.
  Arms: Manual vitrification
Other: Vitrification with GaviTM system — Two oocytes will be frozen by vitrification. At thawing, the degree of rehydration objectified by the measurement of oocyte surfaces and the appearance of potential lysis will be studied thanks to culture in the embryoscope.
  Arms: Automatic vitrification

SUMMARY:
In the space of a few decades, oocyte cryopreservation has become established in the world of reproductive biology with the authorization of oocyte vitrification. This ultra-fast manual freezing technique (authorised in France since 2011) is mainly used to preserve oocytes in women who have to undergo a treatment that could potentially cause sterility. A clear improvement in survival rates since the early stages of slow freezing has been observed with vitrification but with fairly heterogeneous results Indeed, manual vitrification remains an operator-dependent technique with a long learning curve and which does not allow an oocyte survival rate of more than 70-80%.

The recent marketing of an automatic vitrification machine would make it possible to standardise the whole vitrification process from the contact/exchange of fluids to the sealing of the units, and thus potentially increase the oocyte survival rate. It seems to be in the best interest of women that their ability to conceive be preserved (probably for several years) with the technique that offers the best survival and reproducibility rates.

However, no studies have been conducted to assess the impact of such automation on oocyte survival.

For this reason the investigators wish to set up a comparative study between the routine, manual technique, and an automated technique (GAVI system), using immature oocytes, not suitable for fertilization, and usually discarded.

ELIGIBILITY:
Inclusion Criteria:

Patient must be:

* Adult
* Affiliated to a National Health System
* Informed about the study and having given consent
* Receiving an in vitro fertilization attempt with microinjection (ICSI, IntraCytoplasmic Sperm Injection) or having agreed to donate oocytes after approval by the Multidisciplinary Committee
* Having more than two immature, non-fertile oocytes on the day the oocytes are retrieved,
* Having at least two mature oocytes at the end of a 24-hour maturation in vitro.

Exclusion Criteria:

* Protected patient, under guardianship or trusteeship
* In Vitro Fertilization (IVF) Attempts
* Attempts at IVF or ICSI performed in the context of viral risk (both systems will be frozen in the same nitrogen tanks in the assisted reproduction laboratory)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2018-01-01 (Actual); Primary Completion 2020-08 (Estimated); Study Completion 2020-08 (Estimated)

PRIMARY OUTCOMES:
absence of post-thaw oocyte lysis | At warming
absence of post-thaw oocyte lysis | 3 hours after warming

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Dijon Bourgogne, Dijon, France

REFERENCES:
- [Derived] Barberet J, Ducreux B, Bruno C, Guilleman M, Simonot R, Lieury N, Guilloteau A, Bourc'his D, Fauque P. Comparison of oocyte vitrification using a semi-automated or a manual closed system in human siblings: survival and transcriptomic analyses. J Ovarian Res. 2022 Dec 5;15(1):128. doi: 10.1186/s13048-022-01064-3. PMID 36464714